CLINICAL TRIAL: NCT07396779
Title: The Effects of Cognitive Task-Based Walking Exercise on Cognitive Function, Depression, Sleep Quality, and Quality of Life in Older Adults With Brain Fog: A Randomized Controlled Trial
Brief Title: Cognitive Task-Based Walking Effects on Cognition, Mood, Sleep, and Quality of Life in Older Adults With Brain Fog
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre DANSUK, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7890
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Brain Fog; Cognitive Impairment; Geriatric Population
Keywords: Brain Fog; Cognitive Task-Based Exercise; Walking Exercise; Cognitive Function; Sleep Quality; Quality of Life
MeSH Terms: conditions — Mental Fatigue; Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study is a single-center, prospective, randomized controlled trial comparing cognitive task-based walking exercise with walking-only exercise in older adults with brain fog. Participants will undergo supervised low-intensity walking exercises three times per week for four weeks. Outcomes will be evaluated at baseline and post-intervention to determine the effects on cognitive function, depression, sleep quality, and quality of life.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to group allocation. Participants will not be informed whether they are assigned to the cognitive task-based walking exercise group or the walking-only exercise group. Outcome assessors will be independent from the intervention process and will be unaware of group assignments during baseline and post-intervention assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Task-Based Walking Exercise (Experimental): Participants will perform low-intensity walking exercises combined with concurrent cognitive tasks under physiotherapist supervision, three times per week for four weeks.
  Interventions: Other: Cognitive Task-Based Walking Exercise
- Walking-Only Exercise (Active Comparator): Participants will perform the same low-intensity walking exercise protocol without cognitive tasks, under physiotherapist supervision, three times per week for four weeks.
  Interventions: Other: Walking-Only Exercise

INTERVENTIONS:
Other: Cognitive Task-Based Walking Exercise — Participants will perform supervised low-intensity walking exercises combined with concurrent cognitive tasks targeting attention, memory, and executive functions. Exercise sessions will be conducted three times per week for four weeks under the supervision of a physiotherapist.
  Arms: Cognitive Task-Based Walking Exercise
Other: Walking-Only Exercise — Participants will perform supervised low-intensity walking exercises without concurrent cognitive tasks. Exercise sessions will be conducted three times per week for four weeks under the supervision of a physiotherapist.
  Arms: Walking-Only Exercise

SUMMARY:
This randomized controlled trial aims to investigate the effects of cognitive task-based walking exercise on cognitive function, depressive symptoms, sleep quality, and quality of life in older adults experiencing brain fog. Eligible participants will be randomly assigned to either a cognitive task-based walking exercise group or a walking-only exercise group. The intervention will be conducted under physiotherapist supervision, three times per week for four weeks. Outcome measures will be assessed at baseline and after the intervention period to compare the effectiveness of the two exercise approaches.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized controlled trial designed to evaluate the effects of cognitive task-based walking exercise on cognitive function, depression, sleep quality, and quality of life in older adults experiencing brain fog. The study will be conducted between November 2025 and May 2026 at the Geriatrics Outpatient Clinic of Istanbul Medipol Mega Hospital.

Participants aged 65 years and older who report a subjective decline in attention, concentration, or mental clarity for at least four weeks and who demonstrate moderate or greater brain fog symptoms according to the Turkish version of the Brain Fog Scale will be eligible for inclusion. Only individuals with preserved global cognitive function (Montreal Cognitive Assessment score ≥20) and the ability to walk independently, with or without an assistive device, will be enrolled. Individuals with diagnosed neurological disorders, severe psychiatric conditions, or medical problems that limit physical activity will be excluded.

Eligible participants will be randomly assigned, using a computer-generated randomization sequence, to one of two groups: (1) a cognitive task-based walking exercise group or (2) a walking-only exercise group. Both groups will participate in supervised, low-intensity walking exercise sessions three times per week for four weeks. Exercise intensity and progression will be individualized according to each participant's physical capacity and balance status.

Each exercise session will include a warm-up phase, a main walking phase, and a cool-down phase. Participants in the cognitive task-based walking exercise group will be required to perform concurrent cognitive tasks during walking, including forward and backward counting, verbal fluency tasks, and sequencing of days of the week and months of the year, targeting attention, memory, and executive functions. The walking-only exercise group will follow the same walking protocol without the addition of cognitive tasks.

Outcome assessments will be conducted at baseline and after the four-week intervention period. Primary and secondary outcomes will include brain fog severity, cognitive function, depressive symptoms, sleep quality, and quality of life. All assessments will be performed by independent outcome assessors who are blinded to group allocation.

The findings of this study are expected to provide evidence regarding the clinical effectiveness of integrating cognitive tasks into walking exercise programs and to support holistic rehabilitation strategies in older adults with brain fog.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Self-reported experience of brain fog symptoms (e.g., reduced attention, concentration, or -mental clarity) for at least the past 4 weeks
* Moderate or higher brain fog severity as determined by the Turkish version of the Brain Fog Scale
* Preserved global cognitive function (Montreal Cognitive Assessment score ≥20)
* Ability to walk independently, with or without an assistive device
* Ability to communicate verbally and follow instructions
* No changes in medication and no acute illness within the past 4 weeks
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Diagnosis of neurological disorders such as Alzheimer's disease or stroke
* History of severe neurological or psychiatric disorders
* Medical conditions that contraindicate participation in physical exercise
* Severe visual or hearing impairments that may interfere with assessments or exercise participation
* Inability to comply with or complete the exercise program

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | Baseline and after 4 weeks
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), which evaluates multiple cognitive domains including attention, memory, executive functions, language, and orientation. Higher scores indicate better cognitive performance.

SECONDARY OUTCOMES:
Brain Fog Scale | Baseline and after 4 weeks
  Brain fog severity will be assessed using the Turkish version of the Brain Fog Scale, a self-reported questionnaire evaluating cognitive, physical, and psychological symptoms. Higher scores indicate greater severity of brain fog symptoms.
Geriatric Depression Scale | Baseline and after 4 weeks
  Depressive symptoms will be evaluated using the Geriatric Depression Scale (GDS), a self-reported questionnaire designed to assess depressive symptoms in older adults. Higher scores indicate greater severity of depressive symptoms.
Pittsburgh Sleep Quality Index | Baseline and after 4 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which measures subjective sleep quality and sleep disturbances over the previous month. Higher scores indicate poorer sleep quality.
World Health Organization Quality of Life Instrument-Older Adults Module | Baseline and after 4 weeks
  Quality of life will be assessed using the World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-OLD). Higher scores indicate better perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Dansuk, PhD, Principal Investigator — Medipol University
Locations (1):
- Emre Dansuk, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No